CLINICAL TRIAL: NCT05517317
Title: Autologous Bone Marrow Mononuclear Cell Infusion for Liver Cirrhosis in Children With Biliary Atresia
Brief Title: Autologous BMNC Infusion for Liver Cirrhosis in Children With BA
Acronym: ABMNCBA
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Vinmec Research Institute of Stem Cell and Gene Technology (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: ISC_22_88
Record Dates: First submitted 2022-08-22; First posted 2022-08-26 (Actual); Last update posted 2022-08-26 (Actual); Status verified 2022-08

CONDITIONS: Biliary Atresia
MeSH Terms: conditions — Biliary Atresia

STUDY DESIGN:
Intervention Model Description: Autologous BMMC infusion
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Autologous BMMC infusion (Experimental): One administration of autologous bone marrow mononuclear cells via the hepatic artery
  Interventions: Combination Product: Autologous BMMC transplantation

INTERVENTIONS:
Combination Product: Autologous BMMC transplantation — One administration of autologous bone marrow mononuclear cells via the hepatic artery

SUMMARY:
To evaluate the safety and early outcomes of autologous bone marrow mononuclear cell (BMMNC) infusion for liver cirrhosis due to biliary atresia (BA) after Kasai operation. An open-label clinical trial was performed from January 2015 to December 2021. 12 children with liver cirrhosis due to BA at the time of Kasai or after Kasai were included. Bone marrow was harvested through anterior iliac crest puncture under general anesthesia. Mononuclear cells (MNCs) were isolated by Ficoll gradient centrifugation and then infused into the hepatic artery.

DETAILED DESCRIPTION:
Biliary atresia (BA) is a progressive fibro-obliterative cholangiopathy and a fatal disease. Without surgery, children with BA rarely survive beyond three years of age. The reported prevalence of BA ranges from 1 in 9640 to 1 in 19,500 live births. In the past, most children with a "non-correctable" type of BA died without adequate treatment. Recently, stem cell administration has been applied in adults with liver cirrhosis and has shown promising outcomes. An open-label clinical trial was performed from January 2015 to December 2021. 12 children with liver cirrhosis due to BA at the time of Kasai or after Kasai were included. Bone marrow was harvested through anterior iliac crest puncture under general anesthesia. Mononuclear cells (MNCs) were isolated by Ficoll gradient centrifugation and then infused into the hepatic artery. Serum bilirubin, albumin, alanine aminotransferase, aspartate aminotransferase, gamma-glutamyl transferase, and prothrombin time were monitored at baseline, three months, six months and 12 months after the transplantation. Esophagoscopies and liver biopsies were performed in patients whose parents provided consent. This study aimed to evaluate both safety and hepatic function after BMMNC administration in these children.

ELIGIBILITY:
Inclusion Criteria:

* Children were diagnosed with Liver Cirrhosis Due to biliary atresia after Kasai's operation
* Two months old or older
* Patients with a manifestation of cirrhosis after Kasai's operation: hepatomegaly, congestive splenomegaly, elevated liver enzymes, Esophageal Varices (based on Endoscopic Diagnosis), cirrhosis (based on liver biopsy)

Exclusion Criteria:

* Epilepsy
* Coagulation disorders
* Allergy to anesthetic agents
* Severe health conditions such as cancer, failure of heart, lung, liver or kidney
* Active infections
* Severe psychiatric disorders

Ages: 2 Months to 15 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 12 (Actual)
Dates: Start 2015-01-01 (Actual); Primary Completion 2022-05-30 (Actual); Study Completion 2022-05-30 (Actual)

PRIMARY OUTCOMES:
Adverse events and serious adverse events | up to the 12-month period following treatment
  To assess safety, the number of AEs or SAEs during stem cell administration (72 h) at 1 month, 3 months, 6 months, and 9 months after discharge will be evaluated

SECONDARY OUTCOMES:
The changes in cholestasis | up to the 12-month period following treatment
  Using Total Bilirubin (units: mg/dL) to measure the changes in cholestasis
The changes in Liver function using Aspart transaminase | up to the 12-month period following treatment
  Using AST (Aspart transaminase) (units: U/L) to measure the changes in liver function.
The changes in Liver function using Alanine transaminase | up to the 12-month period following treatment
  Using ALT (Alanine transaminase) (units: U/L) to measure the changes in liver function.
The changes in Liver function using Gamma GT | up to the 12-month period following treatment
  Using GGT (Gamma GT) (units: U/L) to measure the changes in liver function.
The changes in level of cirrhosis | up to the 12-month period following treatment
  Using PELD score (according to the suggestion of The Liver and Intestinal Organ Transplantation Committee in 2009). PELD is calculated based on three indicators: albumin (g/dL), bilirubin (units: mg/dL) and INR (international normalized ratio). Formula: PELD = 10 * (0.48 * ln(Serum Bilirubin) + 1.857 * ln(INR) - 0.687 * ln(Albumin) + (0.436 if patient is less than 1 year old) + (0.667 if patient has growth failure).
  Evaluate the result:
  If PELD <10: good results
  If 10 <PELD <15: average results
  If PELD> 15: bad results
The changes in liver biopsy | up to the 12-month period following treatment
  Liver biopsy is a powerful clinical tool to evaluate the changes in the level of cirrhosis.

CONTACTS AND LOCATIONS:
Overall Officials: Liem Thanh Nguyen, PhD, Principal Investigator — Vinmec Research Institute of Stem Cell and Gene Technology
Locations (1):
- Vinmec Research Institute of Stem Cell and Gene Technology, Hanoi, Vietnam

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Thanh LN, Nguyen HP, Kieu TPT, Duy MN, Ha HTT, Thi HB, Nguyen TQ, Pham HD, Tran TD. Modified Kasai operation combined with autologous bone marrow mononuclear cell infusion for biliary atresia. BMC Surg. 2024 Nov 20;24(1):368. doi: 10.1186/s12893-024-02669-9. PMID 39568009